CLINICAL TRIAL: NCT00849667
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 3 Study to Assess the Efficacy and Safety of Weekly Farletuzumab (MORAb-003) in Combination With Carboplatin and Taxane in Subjects With Platinum-sensitive Ovarian Cancer in First Relapse
Brief Title: Efficacy and Safety of Farletuzumab (MORAb-003) in Combination With Carboplatin and Taxane in Participants With Platinum-sensitive Ovarian Cancer in First Relapse
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Morphotek (Industry)
Collaborators: Eisai Europe Ltd. (United Kingdom) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MORAb003-004; 2008-005872-29 (EudraCT Number)
Record Dates: First submitted 2009-02-13; First posted 2009-02-24 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; relapsed ovarian cancer; Platinum-sensitive Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — farletuzumab; Carboplatin; taxane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Farletuzumab (1.25 mg/kg) (Active Comparator): Participants will receive farletuzumab 1.25 milligram per kilogram (mg/kg) administer as an intravenous (IV) infusion weekly, followed by taxane (paclitaxel [175 milligram per meter square {mg/m^2}] or docetaxel [75 mg/m^2]), administer as IV infusion and followed by carboplatin (to maintain area under curve [AUC] 5-6 milligram per milliliter per minute [mg/mL/minute]), administer as IV infusion, every three weeks, on Day 1 of each 21-day cycle for 6 cycles (combination therapy). Following completion of combination therapy, maintenance treatment with farletuzumab 1.25 mg/kg, administer as IV infusion, weekly is given until disease progression.
  Interventions: Drug: Farletuzumab; Drug: Carboplatin; Drug: Taxane
- Farletuzumab (2.5 mg/kg) (Active Comparator): Participants will receive farletuzumab 2.5 mg/kg administer as an IV infusion weekly, followed by taxane (paclitaxel [175 mg/m^2] or docetaxel [75 mg/m^2]), administer as IV infusion and followed by carboplatin (to maintain AUC 5-6 mg/mL/minute), administer as IV infusion, every three weeks on Day 1 of each 21-day cycle for 6 cycles (combination therapy). Following completion of combination therapy, maintenance treatment with farletuzumab 2.5 mg/kg, administer as IV infusion, weekly is given until disease progression.
  Interventions: Drug: Farletuzumab; Drug: Carboplatin; Drug: Taxane
- Placebo (Placebo Comparator): Participants will receive farletuzumab-matched placebo (0.9 percent [%] saline) administer as an IV infusion weekly, followed by taxane (paclitaxel [175 mg/m^2] or docetaxel [75 mg/m^2]), administer as IV infusion and followed by carboplatin (to maintain AUC 5-6 mg/mL/minute), administer as IV infusion, every three weeks on Day 1 of each 21-day cycle for 6 cycles (combination therapy). Following completion of combination therapy, maintenance treatment with farletuzumab-matched placebo (0.9% saline), administer as IV infusion, weekly is given until disease progression.
  Interventions: Drug: Carboplatin; Drug: Taxane; Drug: Farletuzumab-matched placebo

INTERVENTIONS:
Drug: Farletuzumab — Farletuzumab IV infusion.
  Other Names: MORAb-003
  Arms: Farletuzumab (1.25 mg/kg); Farletuzumab (2.5 mg/kg)
Drug: Carboplatin — Carboplatin IV infusion.
Drug: Taxane — Taxane (Paclitaxel or Docetaxel) IV infusion.
Drug: Farletuzumab-matched placebo — Farletuzumab-matched placebo IV infusion.
  Arms: Placebo

SUMMARY:
This research is being done to find out if Carboplatin and Taxane works better alone or when given with an experimental drug called MORAb-003(farletuzumab) in subjects with first platinum sensitive relapsed ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* A histologically or cytologically confirmed diagnosis of non-mucinous epithelial ovarian cancer including primary peritoneal or fallopian tube malignancies
* Must have measurable disease by CT or MRI scan
* Must have relapsed radiologically with a randomization date within ≥6 and < 24 months of completion of first-line platinum chemotherapy
* Have been treated with debulking surgery and first-line platinum and taxane based chemotherapy.
* Prior bevacizumbab maintenance is allowed. The last dose of bevacizumab must have been at least 30 days before study Day 1. No cytotoxic maintenance therapy (e.g. taxane) or cancer vaccine therapy is allowed.
* Must be a candidate for carboplatin and taxane therapy
* Neurologic function: neuropathy (sensory and motor) ≤CTCAE Grade 1

Exclusion Criteria:

* Subjects who never responded to first-line platinum-based therapy or whose first relapse occurs <6 months or >24 months from the last platinum therapy
* Subjects who have received other therapy to treat their ovarian cancer since relapse
* Known central nervous system (CNS) tumor involvement
* Evidence of other active invasive malignancy requiring treatment in the past 5 years
* Known allergic reaction to a prior monoclonal antibody therapy or have any documented HAHA
* Previous treatment with MORAb-003 (farletuzumab)
* Clinical contraindications to use of a taxane

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2009-04-16 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2013-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (374):
- United States (110):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Oncology Specialties, PC, Huntsville, Alabama
  - Arizona Hematology & Oncology Associates, Phoenix, Arizona
  - St. Joseph's Hospital, Barrow Neurology Clinics, Phoenix, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Providence St. Joseph Medical Center, Burbank, California
  - California Cancer Care, Inc., Greenbrae, California
  - University of California San Diego, La Jolla, California
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Gynecologic Oncology Associates, Newport Beach, California
  - University of California Davis Cancer Center, Sacramento, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Catholic Health Initiatives, Colorado Springs, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Hematology Oncology P.C., Stamford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - University Cancer Institute, Boynton Beach, Florida
  - Gainsville Hematology Oncology Associates, Gainesville, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Jupiter Medical center Physician's Group, Jupiter, Florida
  - Hematology/Oncology Associates, Lake Worth, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Florida Hospital, Orlando, Florida
  - Sarasota Memorial Healthcare System, Sarasota, Florida
  - Gulfcoast Oncology, St. Petersburg, Florida
  - Oncology-Hematology Associates of W. Broward P.A., Tamarac, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kaiser Permanente - Moanalua Medical Center, Honolulu, Hawaii
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - St. Francis Hospital & Health Centers, Indianapolis, Indiana
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - Hematology & Oncology Specialists, Metairie, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - John Hopkins University, Baltimore, Maryland
  - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Barbara Ann Kamanos Cancer Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Hospital Cancer Center, Kearney, Nebraska
  - The Center for Cancer and Hematologic Disease, Camden, New Jersey
  - Hematology-Oncolgy Associates of NNJ-PA, Denville, New Jersey
  - John Theurer Cancer Center at Hackensack University MC, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arena Oncology Associates, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Piedmont Hematology & Oncology, Winston-Salem, North Carolina
  - Catholic Health Initiatives, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Cancer Care Associates, Tulsa, Oklahoma
  - Providence Oncology & Hematology Care, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Oncology Hematology Associates, DuBois, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, PA, Austin, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Baylor Sammons Cancer Center, Dallas, Texas
  - International Beneficence Clinical Research, L.L.C., Harlingen, Texas
  - University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - South Texas Oncology and Hematology, PA, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - US Oncology Research, Wichita Falls, Texas
  - Northern Utah Associates, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - Peninsula Cancer Institute - Riverside Gynecology Oncology, Newport News, Virginia
  - Harrison Bremerton Hematology and Oncology, Bremerton, Washington
  - Providence Everett Medical Center, Everett, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - Aurora Health Care, West Allis, Wisconsin
- Argentina (12):
  - Hospital Zonal Especializado en Oncología de Lanús, Buenos Aires
  - Consultorios Medicos Privados SA, Buenos Aries
  - Fundación Sanatorio Güemes, CABA
  - Clinica Universitaria Reina Fabiola, Códoba
  - Instituto Medico Platense, La Plata
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Hospital Bocalandro, Loma Hermosa
  - Centro Oncologico Integral, Mar del Plata
  - CER Instituto Medico, Quilmes
  - Centro Médico San Roque, San Miguel de Tucumán
  - Centro Medico de Alta Complejidad Cemac, San Salvador de Jujuy
  - ISIS Centro Especializado de LUCE SA, Santa Fe
- Australia (6):
  - Tweed Hospital, Tweed Heads, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - North Adelaide Oncology Clinical Trials, North Adelaide, South Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (3):
  - Kaiser-Franz-Josef Spital, Vienna
  - Krankenhaus Wien-Hietzing, Vienna
  - Landeskrankenhaus Villach, Villach
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge - Campus Maria's Voorzienigheid, Kortrijk
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - Sint-Augustinuskliniek, Wilrijk
- Brazil (21):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Instituto de Pesquisas Clínicas para Estudos Multicêntricos, Caxias do Sul
  - Santa Casa da Misericórdia de Curitiba, Curitiba
  - Instituto do Câncer do Ceará - ICC, Fortaleza
  - Hosp. Araujo Jorge, Goiânia
  - Associação Hospital de Caridade Ijuí, Ijuí
  - Clinica de Neoplasias Litoral, Itajaí
  - Hospital Amaral Carvalho, Jaú
  - Liga Norte-Riograndense Contra o Câncer, Natal
  - Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Clínica de Oncologia de Porto Alegre S/S Ltda, Porto Alegre
  - Instituto Ribeirãopretano de Combate ao Câncer, Ribeirão Preto
  - Clínica Oncologistas Associados, Rio de Janeiro
  - INCA - Instituto Nacional do Câncer, Rio de Janeiro - RJ
  - Hospital Santa Izabel - Santa Casa de Misericordia da Bahia, Salvador
  - Clínica AMO - Assistência Multidiciplinar em Oncologia, Salvador
  - Centro de Estudos de Oncologia da FMABC, Santo André
  - Saúde ABC Serviços Médicos Hospitalares Ltda, Santo André
  - Instituto do Câncer Arnaldo Vieira de Carvalho, São Paulo
  - Certo Oncologia, São Paulo
  - Hospital Premier, São Paulo
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cancer Center For The Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency, Surrey, British Columbia
  - BCCA, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Ottawa Hospital, Ottawa, Ontario
- Chile (3):
  - Instituto de Terapias Oncologicas, Santiago
  - Instituto Clínico Oncológico del Sur, Temuco
  - Instituto Oncologico Ltda., Viña del Mar
- France (5):
  - Centre Régional de lutte contre le cancer Paul Papin, Angers
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint Louis, Paris
  - Institut Jean Godinot - Centre de lutte contre le cancer, Reims
- Germany (17):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Helios Klinikum Berlin-Buch, Buch
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Marien-Hospital Akademisches Lehrkrankenhaus, Düsseldorf
  - Frauenarztpraxis Dr. med. Gröll de Rivera, Ebersberg
  - Universitätsklinikum Essen, Essen
  - Krankenhaus Nordwest, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Kath. Marienkrankenhaus gGmbH, Hamburg
  - Universität Heidelberg, Heidelberg
  - St. Vincentius Kliniken Karlsruhe, Karlsruhe
  - Universitätsklinik Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München - Innenstadt, München
  - Rotkreuzklinikum München, München
  - Klinikum Südstadt Rostock, Rostock
  - Klinikum Traunstein, Traunstein
- Greece (5):
  - University General Hospital of Heraklion, Heraklion, Crete
  - Alexandra Hospital, Athens
  - General Oncology Hospital Kifissias "Oi Agioi Anargyroi", Athens
  - University General Hospital of Patras, Pátrai
  - Papageorgiou General Hospital, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, Pokfulam, Islands District
  - Tuen Mun Hospital, Tuenmen
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Bács-Kiskun Megyei Önkormányzat Kórháza, Kecskemét
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelöintézet, Szolnok
  - Veszprém Megyei Önkormányzat Csolnoky Ferenc Kórház-Rendelöintézet, Veszprém
- India (18):
  - Apollo Hospitals International Limited, Gandhinagar, Gujarat
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Jawaharlal Nehru Cancer Hospital & Research Centre, Bhopal, Madhya Pradesh
  - Jehangir, Clinical Development Centre, Pune, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Dr. Kamakshi Memorial Hospital, Chennai, Tamil Nadu
  - Chittaranjan National Cancer Institute, Kolkata, West Bengal
  - M.S Ramaiah Medical College and Teaching Hospital Ethical Review Board, Bangalore
  - MNJ Institute of Oncology and Regional Cancer Centre, Hyderabaad
  - SK Soni Hospital, Jaipur
  - Bhagwan Mahaveer Cancer Hospital and Research Centre, Jaipur
  - Amrita Institute of Medical Sciences and Research Centre, Kochi
  - Lakeshore Hospital, Kochi
  - Tata Memorial Hospital, Mumbai
  - Curie Manavata Cancer Centre, Nashik
  - Shatabdi Superspeciality Hospital, Nashik
  - All India Institute of Medical Sciences, New Delhi
  - Regional Cancer Centre, Trivandrum
- Israel (10):
  - Rambam Medical Center, Haifa
  - Linn Medical Center, Clalit Health Services, Haifa
  - Wolfson Centre, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assaf Harofe Medical Center, Ẕerifin
- Italy (26):
  - Centro di Riferimento Oncologico, Aviano, Pordenone
  - Azienda Ospedaliera Santi Antonio, Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Centro di Ricerca e Formazione ad Alta Tecnologia nelle Scienze Biomediche, Campobasso
  - Azienda Ospedaliera Cannizzaro, Catania
  - Humanitas Centro Catanese di Oncologia, Catania
  - Azienda Ospedaliera Sant'Anna, Como
  - Ospedale di Faenza, Faenza
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Presidio Ospedaliero Vito Fazzi, Lecce
  - Ospedale Mater Salutis ULSS 21 della regione Veneto, Legnago
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Niguarda Cà Granda, Milan
  - Istituto Nazionale per lo studio e la cura dei tumori "Fondazione Giovanni Pascale", Napoli
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Istituto Oncologico Veneto, Padua
  - Ospedale Santa Maria della Misericordia di Perugia, Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Azienda Policlinico Umberto I, Roma
  - Policlinico Universitario "A. Gemelli", Roma
  - Azienda Ospedaliero-Universitaria di Udine, Udine
- Japan (30):
  - Akashi
  - Amagasaki
  - Chiba
  - Fukuoka
  - Hidaka
  - Hiroshima
  - Kagoshima
  - Kashiwa
  - Kawasaki
  - Kōtoku
  - Kumamoto
  - Kure
  - Kurume
  - Matsuyama
  - Minatoku
  - Morioka
  - Nagoya
  - Nakano
  - Niigata
  - Okayama
  - Osaka
  - Sapporo
  - Sayama
  - Sendai
  - Shinjuku-Ku
  - Sunto-Gun
  - Tsu
  - Tsukuba
  - Yamagata
  - Yonago
- Mexico (3):
  - Union Medica Quirurgica de Colima, Colima
  - Triva Investigaciones Medicas Sociedad Anónima de Capital Variable, Morelia
  - Hospital Regional de Veracruz, Veracruz
- Netherlands (4):
  - VU Medisch Centrum, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Orbis Medisch Centrum, Sittard-Geleen
- Philippines (6):
  - Perpetual Succour Hospital, Cebu City, Cebu
  - Cebu Gynecologic Cancer Care Clinic, Cebu
  - Manila Doctors Hospital, Manila
  - San Juan de Dios Hospital, Pasay
  - St. Luke's Medical Center, Quezon City
  - National Kidney and Transplant Institute, Quezon City
- Poland (12):
  - Bialostockie Centrum Onkologii, Bialystok
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Centrum Onkologii, Instytut im. M. Sklodowskiej-Curie oddzial w Gliwicach, Gliwice
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Zaklad Opieki Zdrowotnej MSWiA z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - Olsztynski Osrodek Onkologiczny "Kopernik" Sp. z o.o., Olsztyn
  - Wielkopolskie Centrum Onkologii, Poznan
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Pozna, Poznan
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3, Rybnik
  - Samodzielny Publiczny Szpital Kliniczny nr 2 PAM w Szczecinie, Szczecin
  - Wojskowy Instytut Medyczny, Warsaw
- Portugal (5):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Português de Oncologia Francisco Gentil, Centro Regional de Oncologia de Coimbra, EPE, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil (IPOLFG, EPE), Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil (IPOPFG, EPE), Porto
  - Hospital de São João, Porto
- Russia (8):
  - Kursk Regional Oncology Centre, Kursk
  - Russian Oncology Research Center named after N.N. Blokhin, Moscow
  - Russian Oncology Research Center, Moscow
  - Moscow Research Oncology Institute n.a. P.A.Gertsen, Moscow
  - Medical Radiology Research Center of RAMS, Obninsk
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Republican Clinical Oncology Center of Bashkortostan Republic Ministry of Healthcare, Ufa
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - KK Women's and Children's Hospital, Singapore
- South Korea (7):
  - National Cancer Center, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Cheil General Hospital & Women's Healthcare Center, Seoul
  - Seoul national univercity hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (15):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Vall D'Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial, Barcelona, Catalonia
  - Hospital de Mataró, Mataró, Catalonia
  - Corporació Sanitaria Parc Taulí, Sabadell, Catalonia
  - Hospital Mutua de Terrassa, Terrassa, Catalonia
  - Fundacion Hospital Alcorcon, Alcorcón, Madrid, Communidad de
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Communidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Communidad de
  - Hospital 12 de Octubre, Madrid, Madrid, Communidad de
  - Hospital General Universitario de Elche, Elche, Valencia
  - Fundación Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clinico San Carlos, Madrid
- Universität Zürich, Zurich, Switzerland
- Taiwan (6):
  - National Cheng Kung University Hosptial, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Ukraine (4):
  - Municipal Institution of Cherkasy Regional Counsil "Cherkasy Regional Oncology Dispensary", Cherkasy
  - Chernivtsi Regional Clinical Oncology Dispansery, Chernivtsi
  - Kiev City Oncology Hospital, Kyiv
  - Volyn Regional Oncology Dispensary, Lutsk
- United Kingdom (13):
  - Belfast City Hospital, Belfast
  - Velindre Hospital, Cardiff
  - University Hospital Coventry, Coventry
  - Ninewells Hospital, Dundee
  - Beatson Oncology Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Royal Marsden Hospital, London
  - Hammersmith Hospital, London
  - Clatterbridge Centre For Oncology, Metropolitan Borough of Wirral
  - Derriford Hospital, Plymouth
  - Poole Hospital NHS Trust, Poole
  - Weston Park Hospital, Sheffield
  - New Cross Hospital, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 274 investigative sites in North America, Europe, Asia Pacific, Latin America, and Japan from 16 April 2009 to 12 April 2013.
Pre-assignment Details: A total of 1100 participants were randomized and enrolled, out of which 1091 participants received study treatment. Study was terminated early due to lack of efficacy based on the results for progression-free survival (PFS).
Groups:
- 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin: Participants received farletuzumab 1.25 milligram per kilogram (mg/kg) as an intravenous (IV) infusion, weekly followed by taxane (paclitaxel [175 milligram per meter square {mg/m^2}] or docetaxel [75 mg/m^2]) as IV infusion and carboplatin dose to achieve area under curve (AUC) 5 or 6 milligram per minute per milliliter (mg/min/mL) (carboplatin dose [milligram {mg}] = Target AUC [mg*min/mL]*glomerular filtration rate [GFR] milliliter per minute [mL/min] + 25), administered as IV infusion on Day 1 of each 21-day cycle for 6 cycles in combination therapy. Following completion of combination therapy, maintenance treatment with farletuzumab 1.25 mg/kg as IV infusion, weekly until disease progression, unacceptable toxicity, intercurrent illness, participant or physician requested discontinuation, or investigator's judgement to discontinue treatment (up to maximum 46 cycles-each cycle 21 days).
- 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin: Participants received farletuzumab 2.5 mg/kg as an IV infusion, weekly followed by taxane (paclitaxel [175 mg/m^2] or docetaxel [75 mg/m^2]) as IV infusion and carboplatin dose to achieve AUC 5 or 6 mg/min/mL (carboplatin dose [mg] = Target AUC [mg*min/mL]*GFR [mL/min] + 25), administered as IV infusion on Day 1 of each 21-day cycle for 6 cycles in combination therapy. Following completion of combination therapy, maintenance treatment with farletuzumab 2.5 mg/kg as IV infusion, weekly until disease progression, unacceptable toxicity, intercurrent illness, participant or physician requested discontinuation, or investigator's judgement to discontinue treatment (up to maximum 46 cycles-each cycle 21 days).
- Placebo Plus Taxane and Carboplatin: Participants received farletuzumab-matched placebo (0.9 percent [%] saline) as an IV infusion, weekly followed by taxane (paclitaxel [175 mg/m^2] or docetaxel [75 mg/m^2]) as IV infusion and carboplatin dose to achieve AUC 5 or 6 mg/min/mL (carboplatin dose [mg] = Target AUC [mg*min/mL]*GFR [mL/min] + 25), administered as IV infusion on Day 1 of each 21-day cycle for 6 cycles in combination therapy. Following completion of combination therapy, maintenance treatment with farletuzumab-matched placebo as IV infusion, weekly until disease progression, unacceptable toxicity, intercurrent illness, participant or physician requested discontinuation, or investigator's judgement to discontinue treatment (up to maximum 46 cycles-each cycle 21 days).
Period: Overall Study
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Started | 370 | 366 | 364
Safety Analysis Set | 376 | 363 | 352
Completed | 0 | 0 | 0
Not Completed | 370 | 366 | 364
Not completed — Withdrawal by Subject | 16 | 33 | 35
Not completed — Lost to Follow-up | 8 | 8 | 8
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Other | 18 | 19 | 18
Not completed — Progressive disease | 119 | 100 | 112
Not completed — Sponsor decision | 208 | 204 | 190
Not completed — Investigator discretion | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants randomly assigned to treatment, according to the treatment assigned by the interactive web or voice response randomization system (IWRS/IVRS).
Groups:
- 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin: Participants received farletuzumab 1.25 mg/kg as an IV infusion, weekly followed by taxane (paclitaxel [175 mg/m^2] or docetaxel [75 mg/m^2]) as IV infusion and carboplatin dose to achieve AUC 5 or 6 mg/min/mL (carboplatin dose [mg] = Target AUC [mg*min/mL]*GFR [mL/min] + 25), administered as IV infusion on Day 1 of each 21-day cycle for 6 cycles in combination therapy. Following completion of combination therapy, maintenance treatment with farletuzumab 1.25 mg/kg as IV infusion, weekly until disease progression, unacceptable toxicity, intercurrent illness, participant or physician requested discontinuation, or investigator's judgement to discontinue treatment (up to maximum 46 cycles-each cycle 21 days).
- Placebo Plus Taxane and Carboplatin: Participants received farletuzumab-matched placebo (0.9% saline) as an IV infusion, weekly followed by taxane (paclitaxel [175 mg/m^2] or docetaxel [75 mg/m^2]) as IV infusion and carboplatin dose to achieve AUC 5 or 6 mg/min/mL (carboplatin dose [mg] = Target AUC [mg*min/mL]*GFR [mL/min] + 25), administered as IV infusion on Day 1 of each 21-day cycle for 6 cycles in combination therapy. Following completion of combination therapy, maintenance treatment with farletuzumab-matched placebo as IV infusion, weekly until disease progression, unacceptable toxicity, intercurrent illness, participant or physician requested discontinuation, or investigator's judgement to discontinue treatment (up to maximum 46 cycles-each cycle 21 days).
- Total: Total of all reporting groups
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin | Total
Number analyzed (Participants) | 370 | 366 | 364 | 1100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (10.35) | 58.3 (10.26) | 59.0 (10.22) | 58.6 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 370 | 366 | 364 | 1100
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 38 | 25 | 97
  Not Hispanic or Latino | 331 | 321 | 331 | 983
  Unknown or Not Reported | 5 | 7 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 85 | 76 | 86 | 247
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Black or African American | 5 | 10 | 1 | 16
  White | 272 | 271 | 268 | 811
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time (in months) from the date of randomization to the date of the first observation of progression based on the independent radiologic assessment (modified response evaluation criteria in solid tumors [RECIST]), or date of death, whatever the cause. As per RECIST, disease progression was defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions. If progression or death was not observed for a participant, the PFS time was censored at the date of the last tumor assessment without evidence of progression before the date of initiation of further antitumor treatment, or the cutoff date (whichever was earlier).
Time Frame: From the date of randomization to the date of first documentation of disease progression, or date of death, whichever occurred first (up to 44 months)
Population: ITT population included all participants randomly assigned to treatment, according to the treatment assigned by the IWRS/IVRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 370 | 366 | 364
months | 9.5 [8.6 to 10.2] | 9.7 [8.8 to 10.4] | 9.0 [8.4 to 9.8]
Statistical Analysis 1: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.4513, Log Rank; One-sided log rank test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.81 to 1.21]
Statistical Analysis 2: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.0761, Log Rank; One-sided log rank test; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.70 to 1.06]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of randomization to the date of death, due to any cause. If death was not observed for a participant, the survival time was censored on the last date the participant was known to be alive or the cutoff date, whichever was earlier.
Time Frame: From the date of randomization until date of death from any cause, or study termination by sponsor, whichever came first (up to 48 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 370 | 366 | 364
months | 28.7 [26.6 to 33.5] | 32.1 [26.7 to 35.0] | 29.1 [25.6 to 30.7]
Statistical Analysis 1: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.4823, Log Rank; One-sided log rank test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.78 to 1.27]
Statistical Analysis 2: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.1616, Log Rank; One-sided log rank test; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.68 to 1.13]

3. Secondary Outcome: Cancer Antigen-125 (CA-125) Progression-Free Survival
Description: CA-125 PFS was defined as the time (in months) from the date of randomization until the date of the first observation of progression based on the Rustin criteria, or date of death, whatever the cause. If progression or death was not observed for a participant, the CA-125 PFS time was censored at the date of the last CA-125 assessment without evidence of progression before the date of initiation of further antitumor treatment or the "primary analysis cut off" date, whichever was earlier. Based on Rustin criteria, progressive disease (PD) was a rise in CA125 since beginning of consolidation or previously normal CA125 that rises to greater than or equal to (>=) 2 multiple (*) ULN with either event documented on two occasions or CA-125 >=2*nadir value with either event documented on two occasions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 370 | 366 | 364
months | 13.2 [11.8 to 14.4] | 18.1 [12.7 to NA] — Here NA signifies that the upper limit of confidence interval (CI) was not estimable due to insufficient number of events. | 12.0 [11.1 to 14.6]
Statistical Analysis 1: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.2938, Log Rank; One-sided log-rank test; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.72 to 1.21]
Statistical Analysis 2: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.0318, Log Rank; One-sided log-rank test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.58 to 1.02]

4. Secondary Outcome: Progression-Free Survival Based on Gynecologic Cancer InterGroup (GCIG) Criteria
Description: PFS using GCIG criteria was defined as time (in months) from date of randomization until date of first observation of progression based on GCIG criteria, or date of death, whatever the cause. If progression or death was not observed for a participant, GCIG PFS time was censored at later date of last tumor assessment or CA-125 assessment without evidence of progression before date of initiation of further antitumor treatment or the "primary analysis cut off" date, whichever was earlier. Disease progression per GCIG: Participants with elevated CA-125 pretreatment and normalisation of CA-125 must show evidence of CA-125 >=two times ULN on two occasions at least one week apart or participants with elevated CA-125 pretreatment, which never normalises must show evidence of CA-125 >=two times nadir value on two occasions at least one week apart or participants with CA-125 in normal range pretreatment must show evidence of CA-125 >=two times ULN on two occasions at least one week apart.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 370 | 366 | 364
months | 8.8 [8.4 to 9.7] | 8.6 [8.3 to 9.5] | 8.4 [8.2 to 9.0]
Statistical Analysis 1: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.5636, Log Rank; One-sided log-rank test; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.85 to 1.21]
Statistical Analysis 2: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.1560, Log Rank; One-sided log-rank test; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.76 to 1.09]

5. Secondary Outcome: Percentage of Participants With Length of Second Remission Greater Than First Remission
Description: Length of first remission was defined as a.) the period of time (in months) from the date of completion of previous platinum-based chemotherapy until date of first relapse (that is, first observation of progression). It was assumed that the date of first relapse was the earlier of progression by CA-125 or progression by radiologic assessment, as judged by the investigator using GCIG criteria. b.) the period of time (in months) from the date of completion of previous platinum-based chemotherapy (used prior to study entry) until date of randomization. The length of the second remission was defined as the period of time (in months) from the date of completion of platinum-based chemotherapy until the first observation of progression based on GCIG criteria. Based on GCIG criteria, disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions.
Time Frame: From the date of last dose of platinum-based chemotherapy to date of relapse and date of last dose of platinum-based chemotherapy to first observation of progression (up to 48 months)
Population: ITT population included all participants randomly assigned to treatment, according to the treatment assigned by the IWRS/IVRS. Here "N" overall number of participants analyzed included all participants with potential for second remission greater than first remission.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 198 | 200 | 201
percentage of participants | 4.0 [1.8 to 7.8] | 6.5 [3.5 to 10.9] | 4.5 [2.1 to 8.3]

6. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response was defined as either a confirmed complete response (CR) or confirmed partial response (PR) as assessed by investigator based on response evaluation criteria in solid tumors version 1.1 (RECIST version 1.1). CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization to the date of first documentation of disease progression, or date of death, whichever occurred first (up to 48 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 370 | 366 | 364
percentage of participants | 57.6 [52.4 to 62.7] | 58.2 [53.0 to 63.3] | 55.8 [50.5 to 60.9]
Statistical Analysis 1: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.6864, Cochran-Mantel-Haenszel; Difference in percentage = 1.8, 95% CI 2-sided [-5.4 to 9.0]
Statistical Analysis 2: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Test type: Superiority; p = 0.4923, Cochran-Mantel-Haenszel; Difference in percentage = 2.4, 95% CI 2-sided [-4.8 to 9.6]

7. Secondary Outcome: Duration of Tumor Response
Description: Duration of response was defined as the time (in months) from first documentation of objective response (confirmed CR or PR) to the first documentation of objective tumor progression or death due to any cause. Duration of response was derived only for those participants with objective evidence of confirmed CR or PR.
Time Frame: From the first date of confirmed objective response (CR or PR) to first date of progression or death due to any cause (up to 48 months)
Population: Analysis performed on a subset of participants who had objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 211 | 211 | 200
months | 8.0 [7.6 to 9.2] | 8.9 [7.7 to 9.7] | 7.6 [7.1 to 8.7]

8. Secondary Outcome: Time to Tumor Response (TTR)
Description: Time to tumor response was defined as the time (in months) from the date of randomization to first documentation of objective tumor response. Time to tumor response was derived for those participants with objective evidence of CR or PR.
Time Frame: From the date of randomization to first documentation of objective response (up to 48 months)
Population: Analysis performed on a subset of participants who had objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 211 | 211 | 200
months | 1.5 [1.4 to 1.7] | 1.5 [1.4 to 1.7] | 1.5 [1.4 to 1.9]

9. Secondary Outcome: Percentage of Participants With Serologic Response (SR)
Description: SR was defined as either normalization, 75% response, or 50% response using the Rustin criteria. Percentage of participants with 50% SR, 75% SR and SR leading to normalization were reported. A 50% response according to CA-125 was defined as a 50% decrease in serum CA-125 levels, as determined through a series of four CA-125 samples (one baseline sample with an elevated level, the sample that showed a 50% decrease, and a confirmatory sample at the decreased level). A 75% response was established if there had a serial decrease in serum CA-125 levels of 75% over three samples. In both the 50% and 75% response definitions, the final sample was analyzed at least 28 days after the previous sample.
Time Frame: Up to 48 months
Population: SR Evaluable Populations included all randomized participants who received at least one dose of study drug and who had a baseline and at least one assessment during treatment, sufficient to assess the endpoint of interest.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 273 | 273 | 272
percentage of participants
  50% SR (Responder) | 91.9 [88.1 to 94.9] | 97.4 [94.8 to 99.0] | 92.3 [88.4 to 95.2]
  75% SR (Responder) | 86.1 [81.4 to 90.0] | 85.7 [81.0 to 89.6] | 82.0 [76.9 to 86.4]
  SR leading to normalization (Responder) | 65.2 [59.2 to 70.8] | 64.8 [58.9 to 70.5] | 59.9 [53.8 to 65.8]
Statistical Analysis 1: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; 50% serological response; Test type: Superiority; p = 0.8106, Cochran-Mantel-Haenszel; Difference in percentage = -0.4, 95% CI 2-sided [-4.9 to 4.1]
Statistical Analysis 2: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; 50% serological response; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel; Difference in percentage = 5.1, 95% CI 2-sided [1.4 to 8.8]
Statistical Analysis 3: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; 75% serological response; Test type: Superiority; p = 0.3005, Cochran-Mantel-Haenszel; Difference in percentage = 4.1, 95% CI 2-sided [-2.0 to 10.2]
Statistical Analysis 4: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; 75% serological response; Test type: Superiority; p = 0.2445, Cochran-Mantel-Haenszel; Difference in percentage = 3.7, 95% CI 2-sided [-2.5 to 9.9]
Statistical Analysis 5: Comparison: 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Serologic response leading to normalization; Test type: Superiority; p = 0.2797, Cochran-Mantel-Haenszel; Difference in percentage = 5.3, 95% CI 2-sided [-2.8 to 13.4]
Statistical Analysis 6: Comparison: 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin vs Placebo Plus Taxane and Carboplatin; Serologic response leading to normalization; Test type: Superiority; p = 0.2136, Cochran-Mantel-Haenszel; Difference in percentage = 4.9, 95% CI 2-sided [-3.2 to 13.0]

10. Secondary Outcome: Duration of 50% Serologic Response
Description: Duration of SR was defined as the time (in months) from first documentation of response to the first documentation of 50% serologic progression or death due to any cause. For responding participants who did not have serologic progression or did not die and who 1) were either still on study at the time of an analysis, 2) were given antitumor treatment other than study treatment, or 3) were withdrawn from study follow-up before documentation of serologic progression, the duration of SR was censored at the last date the participant was known to be without serologic progression. A 50% response according to CA-125 was defined as a 50% decrease in serum CA-125 levels, as determined through a series of three CA-125 samples (one baseline sample with an elevated level, the sample that showed a 50% decrease, and a confirmatory sample at the decreased level).
Time Frame: From the first date of documentation of response to first documentation of serologic progression or death due to any cause (up to 48 months)
Population: Analysis was performed on a subset of participants who had serologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 251 | 266 | 251
months | 10.7 [9.7 to 12.0] | 12.0 [10.4 to 16.7] | 9.9 [9.0 to 11.5]

11. Secondary Outcome: Time to 50% Serologic Response (TSR)
Description: TSR was defined as the time (in months) from the date of randomization to first documentation of 50% SR. A 50% response according to CA-125 was defined as a 50% decrease in serum CA-125 levels, as determined through a series of three CA-125 samples (one baseline sample with an elevated level, the sample that showed a 50% decrease, and a confirmatory sample at the decreased level).
Time Frame: From the date of randomization to first documentation of 50% SR (up to 48 months)
Population: Analysis was performed on a subset of participants who had serologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 251 | 266 | 251
months | 1.0 [0.9 to 1.0] | 0.9 [0.9 to 1.0] | 1.2 [1.0 to 1.4]

12. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit was defined as a confirmed CR or a confirmed PR, or stable disease (SD) using RECIST 1.0 criteria. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR was defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference smallest sum of longest dimensions since treatment started associated to non-progressive disease response for non target lesions.
Time Frame: Up to 48 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 370 | 366 | 364
percentage of participants | 68.9 | 66.4 | 64.6

13. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration of Total Carboplatin and Total Paclitaxel
Time Frame: Cycle 2 Week 1 Day 1: 0-45 hours post-dose (cycle length=21 days)
Population: Pharmacokinetic Analysis Set included all participants who have sufficient pharmacokinetic data to derive at least one pharmacokinetic parameter. Here "overall number of participants analyzed" signifies participants who were analyzed for this outcome measure. Pharmacokinetic data was collected and analyzed only for a maximum of 7 participants in this study.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 1 | 2 | 4
microgram per milliliter (mcg/mL)
  Total Carboplatin | 19.30 (NA) — Here NA signifies that standard deviation could not be determined because only one participant was analyzed. | 43.55 (22.84) | 21.72 (12.08)
  Total Paclitaxel | 3.29 (NA) — Here NA signifies that standard deviation could not be determined because only one participant was analyzed. | 3.86 (0.20) | 4.95 (2.73)

14. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of Total Carboplatin and Total Paclitaxel
Time Frame: Cycle 2 Week 1 Day 1: 0-45 hours post-dose (cycle length=21 days)
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 1 | 2 | 4
hours
  Total Carboplatin | 0.75 [0.75 to 0.75] | 0.79 [0.50 to 1.08] | 1.96 [0.75 to 3.83]
  Total Paclitaxel | 3.00 [3.00 to 3.00] | 3.21 [3.00 to 3.42] | 3.00 [2.00 to 3.17]

15. Secondary Outcome: AUC (0-inf): Area Under the Concentration-time Curve From Zero (Pre-dose) Extrapolated to Infinite Time of Total Carboplatin and Total Paclitaxel
Time Frame: Cycle 2 Week 1 Day 1: 0-45 hours post-dose (cycle length=21 days)
Population: Pharmacokinetic Analysis Set included all participants who have sufficient pharmacokinetic data to derive at least one pharmacokinetic parameter. Pharmacokinetic data was collected and analyzed only for a maximum of 7 participants in this study. Here "overall number of participants analyzed" signifies participants who were analyzed for this outcome measure. Here "number of participants analyzed" signifies participants who were analyzed for this outcome measure for given categories.
Measure: Mean (Standard Deviation); unit: microgram hour per liter (mcg*h/L)
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 1 | 2 | 3
microgram hour per liter (mcg*h/L)
  Total Carboplatin | 58.70 (NA) — Here NA signifies that standard deviation could not be determined because only one participant was analyzed. | 77.05 (8.41) | 70.37 (10.40)
  Total Paclitaxel: number analyzed (Participants) | 0 | 2 | 3
  Total Paclitaxel |  | 12.30 (1.27) | 16.19 (6.41)

16. Secondary Outcome: T1/2: Terminal Half-life of Total Carboplatin and Total Paclitaxel
Time Frame: Cycle 2 Week 1 Day 1: 0-45 hours post-dose (cycle length=21 days)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 1 | 2 | 4
hours
  Total Carboplatin | 2.94 (NA) — Here NA signifies that standard deviation could not be determined because only one participant was analyzed. | 1.64 (0.31) | 1.72 (0.65)
  Total Paclitaxel: number analyzed (Participants) | 1 | 2 | 3
  Total Paclitaxel | 1.55 (NA) — Here NA signifies that standard deviation could not be determined because only one participant was analyzed. | 4.82 (2.88) | 4.78 (3.24)

17. Secondary Outcome: CL: Clearance of Total Carboplatin and Total Paclitaxel
Time Frame: Cycle 2 Week 1 Day 1: 0-45 hours post-dose (cycle length=21 days)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 1 | 2 | 3
liter per hour (L/h)
  Total Carboplatin | 6.65 (NA) — Here NA signifies that standard deviation could not be determined because only one participant was analyzed. | 8.77 (2.02) | 7.21 (2.40)
  Total Paclitaxel: number analyzed (Participants) | 0 | 2 | 3
  Total Paclitaxel |  | 24.80 (1.27) | 21.00 (11.08)

18. Secondary Outcome: Vd: Volume of Distribution of Total Carboplatin and Total Paclitaxel
Time Frame: Cycle 2 Week 1 Day 1: 0-45 hours post-dose (cycle length=21 days)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 1 | 2 | 3
liter
  Total Carboplatin | 28.20 (NA) — Here NA signifies that standard deviation could not be determined because only one participant was analyzed. | 20.30 (0.85) | 14.86 (5.51)
  Total Paclitaxel: number analyzed (Participants) | 0 | 2 | 3
  Total Paclitaxel |  | 169.50 (94.05) | 110.23 (52.34)

19. Secondary Outcome: Mean Functional Assessment of Cancer Therapy-Ovarian Treatment Outcome Index (FACT-O TOI) Scores
Description: Participant-reported Quality of Life (QoL) was measured using the Functional Assessment of Cancer Therapy-Ovarian (FACT-O), version 4 and reported in the Treatment Outcome Index (TOI) format. TOI is a 26-item subset of the FACT-O questionnaire composed of the raw sum of the physical well-being subscale (7 items), the functional well-being subscale (7 items), and the ovarian cancer subscale (12 items). Each item was scored on a scale of 0 (not at all) to 4 (very much). Some items were reversed scored. Scores from each subsection were summed into one composite score, termed the FACT-O TOI score which ranged from 0 to 104 and a higher score reflected better QoL. As per planned analysis, farletuzumab treatment groups 1.25 mg/kg and 2.5 mg/kg were pooled for the QoL assessment.
Time Frame: Cycle 3, Cycle 6, Cycle 12 (each cycle length=21 days)
Population: The population comprised of all evaluable participants who received at least one dose of farletuzumab or placebo, with study treatment assignment designated according to the IWRS/IVRS, and who completed a baseline FACT-O assessment and at least one follow-up FACT-O assessment during the study. Here "overall number of participants analyzed" signifies participants who were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: Farletuzumab: Participants received farletuzumab 1.25 or 2.5 mg/kg as an IV infusion, weekly followed by taxane (paclitaxel [175 mg/m^2] or docetaxel [75 mg/m^2]) as IV infusion and carboplatin dose to achieve at AUC 5 or 6 mg/min/mL (carboplatin dose [mg] = Target AUC (mg*min/mL)*(GFR [mL/min] + 25), administered as IV infusion on Day 1 of each 21-day cycle for 6 cycles in combination therapy. Following completion of combination therapy, maintenance treatment with farletuzumab 1.25 mg/kg as IV infusion, weekly until disease progression, unacceptable toxicity, intercurrent illness, participant or physician requested discontinuation, or investigator's judgement to discontinue treatment (up to maximum 46 cycles-each cycle 21 days).
Arm/Group | All Participants: Farletuzumab | Placebo Plus Taxane and Carboplatin
Number analyzed (Participants) | 644 | 300
score on a scale
  Cycle 3 | 69.6 (1.0) | 70.7 (1.1)
  Cycle 6 | 70.1 (1.0) | 70.7 (1.1)
  Cycle 12 | 76.2 (1.7) | 72.9 (2.4)

ADVERSE EVENTS:
Time Frame: Up to 48 months
Arm/Group | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin | Placebo Plus Taxane and Carboplatin
All-Cause Mortality (participants affected / at risk) | 143/376 | 119/363 | 121/352
Serious Adverse Events (participants affected / at risk) | 140/376 | 130/363 | 112/352
Other Adverse Events (participants affected / at risk) | 373/376 | 358/363 | 347/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin (N=376) | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin (N=363) | Placebo Plus Taxane and Carboplatin (N=352)
Neutropenia (Blood and lymphatic system disorders) | 35 (43) | 22 (42) | 23 (33)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (18) | 26 (30) | 15 (15)
Anaemia (Blood and lymphatic system disorders) | 14 (18) | 13 (16) | 10 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (14) | 7 (8) | 6 (7)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 10 (10) | 7 (7)
Vomiting (Gastrointestinal disorders) | 10 (11) | 6 (7) | 8 (10)
Ascites (Gastrointestinal disorders) | 7 (10) | 5 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 7 (7) | 8 (9)
Intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 4 (7) | 5 (5)
Ileus (Gastrointestinal disorders) | 5 (7) | 3 (3) | 3 (3)
Small intestine obstruction (Gastrointestinal disorders) | 4 (13) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 7 (7)
Subileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (6) | 5 (5) | 6 (6)
Fatigue (General disorders) | 3 (3) | 3 (3) | 6 (6)
Disease progression (General disorders) | 1 (1) | 2 (2) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0) | 4 (4)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 7 (7) | 6 (6) | 3 (4)
Pneumonia (Infections and infestations) | 3 (3) | 5 (5) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (6) | 3 (3) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 3 (4)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pulmomary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 3 (3)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (3) | 3 (3) | 2 (2)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Colonic Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric Hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric Panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 1 (1) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Catheter Site Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-Organ Disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Ampulla Of Vater Stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 1 (1) | 2 (3)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal Abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Clostridial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Escherichia Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected Lymphocele (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psoas Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster Oticus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective Exacerbation Of Bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia Cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
C-Reactive Protein Increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Magnesium Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Chest X-Ray Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Clostridium Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases To Adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases To Spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Guillain-Barre Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Petit Mal Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Vein Thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urogenital Haemorrhage (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 1 (1)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 2 (2)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obliterative Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Malignant Tumour Excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Mass Excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Ureteral Stent Insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cytoreductive Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Vena Cava Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.25 mg/kg Farletuzumab Plus Taxane and Carboplatin (N=376) | 2.5 mg/kg Farletuzumab Plus Taxane and Carboplatin (N=363) | Placebo Plus Taxane and Carboplatin (N=352)
Nausea (Gastrointestinal disorders) | 215 (486) | 185 (395) | 188 (459)
Diarrhoea (Gastrointestinal disorders) | 134 (251) | 125 (207) | 126 (262)
Vomiting (Gastrointestinal disorders) | 129 (224) | 110 (167) | 103 (211)
Constipation (Gastrointestinal disorders) | 119 (167) | 106 (164) | 101 (155)
Abdominal pain (Gastrointestinal disorders) | 106 (155) | 84 (122) | 91 (149)
Abdominal pain upper (Gastrointestinal disorders) | 46 (55) | 47 (54) | 41 (51)
Dyspepsia (Gastrointestinal disorders) | 44 (57) | 35 (46) | 34 (47)
Stomatitis (Gastrointestinal disorders) | 36 (52) | 25 (28) | 33 (58)
Abdominal distension (Gastrointestinal disorders) | 27 (28) | 25 (29) | 24 (30)
Neutropenia (Blood and lymphatic system disorders) | 205 (622) | 185 (584) | 169 (639)
Anaemia (Blood and lymphatic system disorders) | 139 (214) | 154 (265) | 120 (193)
Thrombocytopenia (Blood and lymphatic system disorders) | 126 (351) | 121 (296) | 99 (237)
Leukopenia (Blood and lymphatic system disorders) | 74 (283) | 72 (194) | 74 (282)
Lymphopenia (Blood and lymphatic system disorders) | 21 (63) | 15 (39) | 21 (85)
Fatigue (General disorders) | 171 (319) | 135 (206) | 149 (319)
Asthenia (General disorders) | 76 (162) | 84 (174) | 64 (134)
Pyrexia (General disorders) | 58 (92) | 47 (67) | 48 (73)
Oedema peripheral (General disorders) | 43 (98) | 37 (43) | 40 (49)
Pain (General disorders) | 32 (43) | 26 (31) | 19 (24)
Mucosal inflammation (General disorders) | 31 (37) | 24 (28) | 30 (51)
Alopecia (Skin and subcutaneous tissue disorders) | 221 (225) | 184 (186) | 202 (207)
Rash (Skin and subcutaneous tissue disorders) | 49 (60) | 40 (52) | 39 (77)
Pruritus (Skin and subcutaneous tissue disorders) | 52 (93) | 36 (56) | 37 (66)
Peripheral sensory neuropathy (Nervous system disorders) | 89 (138) | 71 (117) | 90 (121)
Headache (Nervous system disorders) | 79 (125) | 79 (131) | 71 (137)
Dizziness (Nervous system disorders) | 65 (80) | 52 (69) | 37 (53)
Dysgeusia (Nervous system disorders) | 53 (69) | 51 (65) | 52 (87)
Neuropathy peripheral (Nervous system disorders) | 37 (47) | 44 (53) | 40 (49)
Paraesthesia (Nervous system disorders) | 26 (55) | 24 (48) | 28 (54)
Hypoaesthesia (Nervous system disorders) | 23 (34) | 16 (30) | 12 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 93 (193) | 66 (123) | 86 (170)
Myaligia (Musculoskeletal and connective tissue disorders) | 68 (116) | 63 (95) | 54 (108)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 52 (69) | 48 (72) | 47 (63)
Back pain (Musculoskeletal and connective tissue disorders) | 58 (80) | 30 (34) | 50 (70)
Bone pain (Musculoskeletal and connective tissue disorders) | 24 (26) | 27 (34) | 32 (55)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 (21) | 16 (23) | 25 (29)
Decreased appetite (Metabolism and nutrition disorders) | 95 (195) | 74 (137) | 70 (167)
Hypomagnesaemia (Metabolism and nutrition disorders) | 33 (55) | 33 (42) | 26 (32)
Hypokalaemia (Metabolism and nutrition disorders) | 29 (54) | 34 (54) | 20 (31)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (29) | 21 (26) | 13 (15)
Dehydration (Metabolism and nutrition disorders) | 19 (25) | 15 (21) | 19 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 77 (101) | 61 (84) | 56 (66)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 (60) | 53 (67) | 35 (47)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 25 (27) | 24 (30)
Urinary tract infection (Infections and infestations) | 48 (65) | 41 (66) | 34 (48)
Upper respiratory tract infection (Infections and infestations) | 38 (45) | 38 (59) | 28 (35)
Nasopharyngitis (Infections and infestations) | 46 (63) | 28 (35) | 41 (64)
Insomnia (Psychiatric disorders) | 47 (61) | 39 (41) | 44 (62)
Anxiety (Psychiatric disorders) | 24 (28) | 29 (31) | 15 (15)
Flushing (Vascular disorders) | 25 (34) | 19 (36) | 22 (29)
Hypotension (Vascular disorders) | 21 (24) | 12 (16) | 14 (16)
Hot flush (Vascular disorders) | 16 (29) | 16 (17) | 21 (38)
Drug hypersensitivity (Immune system disorders) | 41 (60) | 52 (94) | 53 (91)
Lacrimation increased (Eye disorders) | 20 (22) | 10 (10) | 8 (8)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 19 (21) | 16 (18) | 19 (22)
FLATULENCE (Gastrointestinal disorders) | 20 (24) | 20 (20) | 17 (20)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 22 (23) | 26 (29) | 20 (24)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 16 (17) | 19 (20) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 (30) | 18 (19) | 15 (21)
Cystitis (Infections and infestations) | 12 (14) | 5 (6) | 19 (23)
Depression (Psychiatric disorders) | 26 (26) | 18 (19) | 8 (8)
Hypertension (Vascular disorders) | 12 (19) | 14 (22) | 19 (22)
Weight decreased (Investigations) | 15 (21) | 19 (19) | 14 (17)
Dysuria (Renal and urinary disorders) | 23 (25) | 20 (23) | 16 (20)

LIMITATIONS AND CAVEATS:
Study termination was based on the primary analysis results for progression-free survival (PFS). Data collection and analyses of health care resource utilization were not performed due to the study being terminated early. Pharmacokinetic data was collected and analyzed for a maximum of only 7 participants in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other